CLINICAL TRIAL: NCT02499887
Title: Repeat Emergency Department Visits Among Patients With Asthma and COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Exclusion criteria prevented enrollment of adequate # of participants
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Heather Lindstrom, Research Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 754754
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone; Albuterol; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care: 30 day albuterol inhaler plus non-tapering course of oral prednisone (50 mg/d) for 4 days (1st dose will have been given in the ED)
  Spacers will be dispensed with all multiple dose inhalers (MDI) to promote proper use and administration of inhaled medications.
  Interventions: Drug: albuterol; Drug: Prednisone
- Treatment (Experimental): Treatment: 30 day QVAR® (beclamethasone dipropionate) inhaler (80 mcg, 1 puff twice daily) plus 30 day albuterol inhaler plus non-tapering course of oral prednisone (50 mg/d) for 5 days
  Spacers will be dispensed with all multiple dose inhalers (MDI) to promote proper use and administration of inhaled medications.
  Interventions: Drug: beclamethasone dipropionate; Drug: albuterol; Drug: Prednisone

INTERVENTIONS:
Drug: beclamethasone dipropionate — Inhaler
  Other Names: Qvar
  Arms: Treatment
Drug: albuterol — Inhaler
  Other Names: Ventolin
Drug: Prednisone — Oral corticosteroid

SUMMARY:
The purpose of the proposed study is to determine whether the addition of inhaled corticosteroids to treatment with oral corticosteroids and albuterol would reduce repeat emergency department (ED) visits among patients treated for acute exacerbations of asthma and COPD discharged from the emergency department to home. The investigators hypothesize that patients treated with inhaled corticosteroids in addition to oral corticosteroids and albuterol will have lower rates of 30-day return visits to the emergency department than those patients treated with oral corticosteroids and albuterol only.

ELIGIBILITY:
Inclusion Criteria:

* Treated in the ED at the Erie County Medical Center (ECMC) for acute symptoms of asthma or COPD during the study period
* Patient age ≥ 18 years
* Resident of the City of Buffalo or Erie County
* Discharged to home
* Patient expresses willingness to return to ECMC or own primary care provider for follow-up visits
* Able to provide informed consent
* Able to comprehend English language

Exclusion Criteria:

* Received oral or inhaled corticosteroids in the week before ED presentation
* Presented to the ED primarily for prescription refills
* Complicated comorbid conditions (e.g. renal disease, cardiovascular disease, CHF, HIV)
* Admitted to ECMC or discharged to another facility
* Previously enrolled during a prior visit to the ED during the study period
* For female patients--pregnant or pregnancy status indeterminate
* Antibiotics are prescribed to treat current asthma/COPD exacerbation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Lindstrom, PhD, Principal Investigator — University at Buffalo, Department of Emergency Medicine
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of Care: 30 day albuterol inhaler plus non-tapering course of oral prednisone (50 mg/d) for 4 days (1st dose will have been given in the ED)
  Spacers will be dispensed with all multiple dose inhalers (MDI) to promote proper use and administration of inhaled medications.
  albuterol: Inhaler
  Prednisone: Oral corticosteroid
- Treatment: Treatment: 30 day QVAR® (beclamethasone dipropionate) inhaler (80 mcg, 1 puff twice daily) plus 30 day albuterol inhaler plus non-tapering course of oral prednisone (50 mg/d) for 5 days
  Spacers will be dispensed with all multiple dose inhalers (MDI) to promote proper use and administration of inhaled medications.
  beclamethasone dipropionate: Inhaler
  albuterol: Inhaler
  Prednisone: Oral corticosteroid
Period: Overall Study
Arm/Group | Standard of Care | Treatment
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Treatment | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants] — Age at presentation to emergency department Population: Information on age of all subjects
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 6
    >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] — Age at presentation to emergency department Population: Information on age of all subjects
  years | 55 [45 to 62] | 57 [52 to 61] | 56 [45 to 62]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of all enrolled subjects Population: Sex of all enrolled subjects
  Participants
    Female | 1 | 0 | 1
    Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Return Visit to the ED Within 30 Days of ED Discharge
Description: Subjects' medical records will be reviewed for the 30 day period following ED discharge to determine if they return to the treating ED or another regional ED for treatment of an acute asthma/COPD exacerbation. Regional ED records will be queried by use of data maintained by HEALTHeLINK, our regional health information organization system. This will allow for more complete capture of ED return visits that could be obtained by looking only at a single ED.
Time Frame: 30 days
Population: Study was discontinued due to low enrollment. No 30 day return visit data was collected.
Arm/Group | Standard of Care | Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrolled patients were contacted within 72 hours of ED discharge. Subjects were asked to describe how they were taking study medications and whether or not they were experiencing any side effects of the medication.
Description: Adverse event description does not differ.
Arm/Group | Standard of Care | Treatment
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No